CLINICAL TRIAL: NCT00054769
Title: Diagnostics For AIDS-Related Pediatric TB, Peru
Brief Title: Diagnosing Tuberculosis in HIV Infected Children in Peru
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 1R01AI049139-01A1 (NIH)
Record Dates: First submitted 2003-02-10; First posted 2003-02-11 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2007-07

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; HIV Infections
Keywords: Pediatrics; Polymerase Chain Reaction
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Tuberculosis is a major cause of mortality among AIDS patients in the developing world. The diagnosis of tuberculosis in HIV infected children is complicated by inefficient and expensive tuberculosis tests and vague diagnostic criteria. This study will evaluate the accuracy and efficiency of several different tuberculosis tests that could be used in developing countries.

DETAILED DESCRIPTION:
HIV infection has been shown to increase mortality from tuberculosis (TB) fivefold in parts of Subsaharan Africa. Increasingly, HIV infected children in developing countries are becoming infected with Mycobacterium tuberculosis (Mtb) and dying at an early age. This project will evaluate novel approaches to the diagnosis of AIDS-related pediatric TB in a hyperendemic setting using rapid, cost-effective Mtb culture and susceptibility methods based on direct microscopic observation techniques. This study will utilize alternative noninvasive Mtb tests that are performed on nasopharyngeal aspirates (NPA) and stool. An optional component will assess improved rapid detection of Mtb by a semi-nested polymerase chain reaction assay (N2 PCR), a technique appropriate for regional reference laboratories in developing countries.

Two hundred-sixty children with clinically diagnosed pulmonary TB (including at least 100 HIV infected children) from the Hospital del Nino, Lima, Peru, and 260 age-matched controls will be enrolled in this study. Mtb will be detected in NPAs and stool by new and traditional culture methods and by N2 PCR. Gastric aspirates from children with a clinical diagnosis of TB will also be tested. Children with a positive N2 PCR but without clinical evidence of TB requiring antituberculous therapy will be followed longitudinally.

ELIGIBILITY:
Inclusion Criteria

* Inability to produce sputum sample
* Clinical picture suggestive of pulmonary TB, score > 7 according to the Stegen and Toledo criteria as adapted by WHO

Exclusion Criteria

* Antituberculous therapy

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 760
Dates: Start 2002-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Oberhelman, MD, Principal Investigator — Tulane School of Public Health and Tropical Medicine
Locations (1):
- Instituto de Salud del Nino, Lima, Lima Province, Peru

REFERENCES:
- [Derived] Oberhelman RA, Soto-Castellares G, Gilman RH, Castillo ME, Kolevic L, Delpino T, Saito M, Salazar-Lindo E, Negron E, Montenegro S, Laguna-Torres VA, Maurtua-Neumann P, Datta S, Evans CA. A Controlled Study of Tuberculosis Diagnosis in HIV-Infected and Uninfected Children in Peru. PLoS One. 2015 Apr 30;10(4):e0120915. doi: 10.1371/journal.pone.0120915. eCollection 2015. PMID 25927526
- [Derived] Oberhelman RA, Soto-Castellares G, Gilman RH, Caviedes L, Castillo ME, Kolevic L, Del Pino T, Saito M, Salazar-Lindo E, Negron E, Montenegro S, Laguna-Torres VA, Moore DA, Evans CA. Diagnostic approaches for paediatric tuberculosis by use of different specimen types, culture methods, and PCR: a prospective case-control study. Lancet Infect Dis. 2010 Sep;10(9):612-20. doi: 10.1016/S1473-3099(10)70141-9. Epub 2010 Jul 23. PMID 20656559